CLINICAL TRIAL: NCT06847139
Title: Effect of Zinc Supplementation on Hyperhomocysteinemia Compared to That of Folic Acid in Patients of Chronic Kidney Disease on Hemodialysis-A Randomized Controlled Trial.
Brief Title: Effect of Zinc Supplementation on Hyperhomocysteinemia Compared to Folic Acid in CKD Patient on Hemodialysis
Acronym: CKD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chittagong Medical College (Other)
Responsible Party: Principal Investigator, Zakwan Ullah, RESIDENT, Chittagong Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PG.2024/1072
Record Dates: First submitted 2025-02-21; First posted 2025-02-26 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Chronic Kidney Disease Requiring Hemodialysis
MeSH Terms: interventions — Zinc Sulfate; Folic Acid; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- patient getting zinc sulfate (Experimental): patient will get zinc sulfate 50 mg daily
  Interventions: Drug: Zinc Sulfate 50 Mg Tab
- patient getting folic acid (Active Comparator): patient will get folic acid 5 mg
  Interventions: Drug: Folic Acid 5 Mg Oral Tablet

INTERVENTIONS:
Drug: Zinc Sulfate 50 Mg Tab — experimental group will get zinc sulfate
  Arms: patient getting zinc sulfate
Drug: Folic Acid 5 Mg Oral Tablet — control group will get folic acid
  Arms: patient getting folic acid

SUMMARY:
Hyperhomocysteinemia is a well-recognized risk factor for accelerated cardiovascular events in hemodialysis patients. Hyperhomocysteinemia is common in individuals with chronic kidney disease (CKD). Zinc is a vital cofactor for homocysteine metabolism enzymes. Although numerous studies have demonstrated the efficacy of folic acid in hyperhomocysteinemia, zinc supplementation has the potential to reduce homocysteine levels in hemodialysis patients. Objective: To evaluate the effect of Zinc supplementation on hyperhomocysteinemia compared to that of folic acid in patients with chronic kidney disease on hemodialysis. Materials and Methods: This open-label randomized active-controlled trial will be conducted in the Department of Nephrology of Chittagong Medical College Hospital, Chattogram, Bangladesh, for one and a half years. A total of ninety CKD patients on maintenance hemodialysis will be included in the study. Patients will be randomly divided into two groups. The experimental group will be treated with zinc sulfate (50 mg elemental zinc/day) for six weeks in conjunction with conventional treatment for CKD. The Control group will receive folic acid (5mg/day) along with conventional medications for CKD. The primary outcome measure will be the change in the plasma homocysteine level after 6 weeks, while the other variables will include serum creatinine, eGFR, serum albumin and C-reactive protein (CRP) level. Adverse events and safety measures will also be recorded. The primary analysis will be an intention to treat analysis performed with SPSS-23. Data from previous studies indicate zinc supplementation can reduce homocysteine levels in CKD patients facilitating its metabolism. Additionally, the anti-inflammatory properties of zinc may facilitate homocysteine reduction. Moreover, zinc is crucial in various physiological processes, including immune function, protein synthesis, and wound healing. Further clinical trials are still needed to understand better the safety and efficacy of zinc supplementation in CKD patients.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥18 years 2. Patient with chronic kidney disease on HD for ≥ 3 months 3. Plasma homocysteine level > 15μmol/L

Exclusion Criteria:

1. Acute illness at the time of inclusion.
2. Diagnosed case of malabsorption
3. Planned major surgery
4. Renal transplantation
5. Receiving zinc or folic acid supplementation within the previous month from enrollment.
6. Concomitant use of vitamin B 12 supplementation(6 days), corticosteroid (18-36 hour), anti folate or cytotoxic drugs, quinolones, tetracyclines, bisphosphonates.
7. Known hypersensitivity to zinc or folic acid.

   -

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
change from baseline plasma homocysteine level after intervention | six week

CONTACTS AND LOCATIONS:
Locations (1):
- Chittagong Medical College, Chittagong, Bangladesh